CLINICAL TRIAL: NCT05507034
Title: sCANsens: Identifying Biomarkers for Chronic Pain After Breast Cancer Treatment
Brief Title: Identifying Biomarkers for Chronic Pain After Breast Cancer Treatment.
Acronym: sCANsens
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, Prof. dr. Mira Meeús, Prof. Dr., Universiteit Antwerpen
Other Study IDs: 1780
Record Dates: First submitted 2022-07-05; First posted 2022-08-18 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Neoplasm, Breast; Carcinoma Breast; Chronic Pain
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain | interventions — Environmental Biomarkers; Gene Expression; Polymorphism, Single Nucleotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer: Breast cancer patients following over time during cancer treatment
  Interventions: Diagnostic Test: Biomarkers

INTERVENTIONS:
Diagnostic Test: Biomarkers — Each intervention is performed at 4 timepoints namely: before surgery, i.e. baseline (T0), 1-3 weeks post-surgery (T1), 3 months post-surgery (T2) and 1 year post-surgery (T4)
  Other Names: Questionnaires: Depression Anxiety Stress Scales Short form, Pain Catastrophising Scale, VK+ and Positive and Negative Affect Schedule; Quantitative sensory testing: hyperalgesia using TSA2 (Medoc), Conditioned Pain Modulation using TSA2 (Medoc), Temporal Summation using monofilament (256mN Optihair-2 Set) and TSA2 (Medoc); Brain imaging: T1 MPRAGE, rsfMRI, Diffusion Weighted Image and T2 sequence.; Blood analysis: Cytokine and Brain-Derived Neurotrophic Factor expression measurements, SNPs and CpG methylation detection.

SUMMARY:
Up to 40% of women experience chronic pain after treatment for breast cancer, and this pain is often very disabling. However, chronic pain after breast cancer remains under-recognised and undertreated. An effective and patient-tailored approach of (chronic) pain after breast cancer indeed requires a thorough knowledge and

evaluation of the pain. In daily clinical practice, however, guidelines for a comprehensive diagnosis of pain in cancer patients and survivors are lacking. Further research in this topic is crucial for an efficient, preventive as well as curative, approach of pain after breast cancer. Besides the high prevalence and the important impact of pain in this population, the breast cancer population is also an ideal population to study chronic pain and its natural time course in different stages, since most patients start pain-free, but almost half of them end up

with chronic pain. Therefore, this study aims to map biomarkers (both predictive, prognostic and diagnostic) for chronic pain after breast cancer treatment. We will study possible biopsychosocial biomarkers in

relation to (chronic) pain and monitor their temporal changes from the moment of diagnosis until 1 year after surgery. The potential biomarkers are situated within the medical imaging of the brain, measurements of pain sensitivity and psychological variables.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral breast cancer
* Pain at enrollment <3/10 on average during the past week
* First cancer diagnosis

Exclusion Criteria:

* Pre-existing pain conditions
* major pre-existing neurological disorders
* No recurrent cancer or metastasis
* No previous surgery in area

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagnosed with unilateral breast cancer
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Localisation of pain | Time frame up to 1 year post-surgery
  Localisation and experience of pain after cancer treatment measured with the Mc Gill Pain Questionnaire Dutch Language Version: Anamnesis questions to localize the pain and the experience of the patient. Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
Pain intensity | Time frame up to 1 year post-surgery
  Visual Analogue Scale included in the Mc Gill Pain Questionnaire is a 100mm horizontal line were the patient is asked to indicate his/her perceived pain intensity at this moment, the minimum and the maximum of the pain. Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
Influence of pain on the quality of life | Time frame up to 1 year post-surgery
  Quality of Life questions included in the Mc Gill Pain Questionnaire: self-report to indicate the impact of pain on quality of life. The higher the score the higher the impact (0-27). Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
Severity of pain symptoms | Time frame up to 1 year post-surgery
  Adjective list of pain symptoms included in the Mc Gill Pain Questionnaire Dutch : Language Version (0-63): Self-report of pain evaluating the sensory intensity, emotional impact and the cognitive evaluation of pain. Each part or dimension of the MPQ is individually scored and a cumulative total score is also recorded. Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery

SECONDARY OUTCOMES:
Prognostic value of Pain Catastrophizing | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Pain Catastrophizing Scale (0-52) : It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Prognostic value of Depression, Anxiety and Stress | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Depression, Anxiety and Stress Scale (DASS-21) (range 0-132). The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress
Prognostic value of Positive and Negative affect | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Positive and Negative Affect Schedule (10-50): This scale consists of different words that describe feelings and emotions, it measures positive and negative affect. Lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Prognostic value of Resilience | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  VK+ : This scale gives an indication about the resilience of the patients (0-100). The higher the score, the more resilience is present.
Prognostic value of hyperalgesia | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Cold and hot detection and pain thresholds are measured as the first identified stimulus under increasing stimulus intensities. Thresholds are measured at local places to evaluate primary hyperalgesia and a distant location to assess secondary hyperalgesia. Results are compared with normative data.
Prognostic value of conditioned pain modulation | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  'Test' stimulus and a 'conditioning' stimulus applied is used to assess pain sensitivity to a warmth stimulus pre- and post the noxious conditioning stimulus and the difference is calculated between premeasures and postmeasures. When the second pressure pain threshold (i.e., test stimulus) is similar or lower than the first, dysfunctional inhibitory pain mechanisms are present.
Prognostic value of temporal summation | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Repetitive stimuli are given of which the perceived intensity of the stimulus (first, last and after sensations) is measured by a Numeric Rating Scale. The difference between the first and the last stimuli is calculated in order to determine the temporal summation. Enhanced temporal summation is considered as positive with at least two points of increase on the NRS
Prognostic value of gray matter differences | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  T1 acquisition and Voxel-Based Morphometry is used to measure regional differences in gray matter. T2 acquisition is applied for possible co-registration and improving robustness for post-processing pipelines.
Prognostic value of functional connectivity | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Rs-fMRI acquisition is used to measure functional connectivity.
Prognostic value of Fractional Anisotropy | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Diffusion Weighted Imaging acquisition is used to assess differences in fractional anisotropy. T2 acquisition is applied for possible co-registration and improving robustness for post-processing pipelines.
Prognostic value of the percentage CpG methylation in gene regions of selected cytokine and Brain Derived Neurotrophic Factor genes. | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Genes associated with the persistent pain phenotype will be selected using multivariate analysis. CpG methylation is determined using bisulfate CpG pyrosequencing. PyroMark Q24 Analyses software will assess the average methylation of each CpG in the different gene regions of interest and return a percentage (from 0-100% methylation) as a result.
Prognostic value of cytokine expression | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Interested cytokines will be selected using multivariate analyses. Plasma samples will be assessed using a multiplex panel.
Prognostic value of Brain Derived Neurotrophic factor expression | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  Measurements of soluble Brain Derived Neurotrophic factor expression is assessed using enzyme-linked immunosorbent assay.
Prognostic value of single nucleotide polymorphisms (SNPs) | Assessment at T0: pre-surgery, T1: 1-3 weeks post-surgery, T2: 3 months post-surgery, T3: 1 year post-surgery
  A total of 82 SNPs from 15 cytokine genes and 2 SNPs of brain derived neurotrophic factor will be analysed using a SNP genotyping assay.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Meeus, Prof., Principal Investigator — Universiteit Antwerpen; An De Groef, Prof., Study Chair — Universiteit Antwerpen
Locations (1):
- University Hospital Antwerpen, Wilrijk, Antwerpen, Belgium

REFERENCES:
- See also: Related Info — https://www.caredon.org/researchers/projects/biomarkers-pain